CLINICAL TRIAL: NCT00607100
Title: High-Resolution Optical Coherence Tomography for Detection of Retinal Nerve Fiber Layer Loss in Band Atrophy of the Optic Nerve
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Mario Luiz Ribeiro Monteiro, Phd, University of São Paulo
Other Study IDs: CAPPESQ N. 1056/07
Record Dates: First submitted 2008-02-04; First posted 2008-02-05 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Band Atrophy; Chiasmal Compression; Neural Loss
Keywords: High-Resolution Optical Coherence Tomography; Retinal Nerve Fiber Layer; Band Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with Band atrophy of the optic nerve
- 2: Normal Controls

SUMMARY:
The purpose of this study is to compare the abilities of high-speed,high-resolution (HR) optical coherence tomography (OCT) and Stratus OCT for detection of retinal nerve fiber layer (RNFL) loss in eyes with band atrophy (BA) of the optic nerve.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity better than 20/30
* Refractive error less 5 spherical diopter and 3 cylinder diopter
* Temporal field defect

Exclusion Criteria:

* Presence of glaucoma and optic nerve anomalies
* A normal nasal field

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with band atrophy from chismal compression and controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-03 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Costa Cunha, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo - Ophthalmology Department, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Costa-Cunha LV, Cunha LP, Malta RF, Monteiro ML. Comparison of Fourier-domain and time-domain optical coherence tomography in the detection of band atrophy of the optic nerve. Am J Ophthalmol. 2009 Jan;147(1):56-63.e2. doi: 10.1016/j.ajo.2008.07.020. Epub 2008 Sep 6. PMID 18774548